CLINICAL TRIAL: NCT05577481
Title: Research on the Efficacy and Brain Network Mechanism of Personalized Targeting Intermittent Theta Burst Stimulation (iTBS) Based on Functional Magnetic Resonance Imaging for the Treatment of Major Depressive Disorder
Brief Title: Neuronavigation Guided iTBS With Personalized Target for Depression
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJLL-KY20222111
Record Dates: First submitted 2022-09-25; First posted 2022-10-13 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-03

CONDITIONS: Depression
Keywords: depression; intermittent Theta Burst Stimulation; neuronavigation
MeSH Terms: conditions — Depression | interventions — Antidepressive Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- functional MRI-guided iTBS(sham group) (Sham Comparator): The stimulating site of the left DLPFC is targeted based on functional MRI, where the most negative functional connectivity with the left pgACC. The MNI coordinate is (-10, 42, 6).
  Interventions: Combination Product: sham iTBS combined with antidepressants
- functional MRI-guided iTBS (pgACC-DLPFC) (Experimental): The stimulating site of the left DLPFC is targeted based on functional MRI, where the most negative functional connectivity with the left pgACC. The MNI coordinate is (-10, 42, 6).
  Interventions: Combination Product: iTBS combined with antidepressants

INTERVENTIONS:
Combination Product: sham iTBS combined with antidepressants — Two sessions of sham prolonged iTBS (1800 pulses) per day over 10 days combined with antidepressants.
  Arms: functional MRI-guided iTBS(sham group)
Combination Product: iTBS combined with antidepressants — Two sessions of prolonged iTBS (1800 pulses) per day over 10 days combined with antidepressants.
  Arms: functional MRI-guided iTBS (pgACC-DLPFC)

SUMMARY:
The study will compare the efficacy of intermittent Theta Burst Stimulation (iTBS) with DLPFC-pgACC personalized target for major depressive disorder (MDD) and explore possible brain network mechanisms. The stimulated targets will be located by magnetic resonance imaging (MRI) based on functional MRI based on functional connectivity respectively. This study aims to identify that functional connectivity targeted iTBS protocols on DLPFC-pgACC personalized target have a better antidepressant efficacy compared the sham group and certify that pgACC is an effective potential effector target.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years old
* Meet the criteria of the Diagnostic and Statistical Manual of Mental Disorder- V of MDD, single or recurrent
* Meet the threshold on the total HAMD17 score of >17 at both screening and baseline visits
* Able to provide informed consent

Exclusion Criteria:

* any other current or past psychiatric axis-I or axis-II disorders
* severe physical illnesses
* psychotic symptoms, alcohol or drug abuse
* A history of neurological disorders including seizure, cerebral trauma
* MRI evidence of structural brain abnormalities
* Contraindications to MRI and rTMS
* Acute suicide
* Female that is pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in the 17-Item Hamilton Rating Scale for Depression (HAMD-17) Score from Baseline to 4 weeks post treatment | baseline and 4-week post treatment
  The HAMD-17 total score comprises a sum of the 17 individual item scores. Each item is rated on a 3 points scale from 0 to 2. The Total Score can range from 0 to 52, and higher scores indicate a greater degree of depression.

SECONDARY OUTCOMES:
Therapeutic response rate and remission rate | immediately post-treatment
  Response is defined as a reduction ≥ 50% on the HAMD-17 and remission is defined as a score <8 on the HAMD-17.
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) Score | baseline, immediately post-treatment and 2-week, 4-week and 8-week post-treatment
  MADRS total score comprises a sum of the 10 individual item scores. Each item is rated on a 7 point scale from 0 to 6. The Total Score can range from 0 to 60, and higher scores indicate a greater degree of depression.
Change in the Beck Scale for Suicidal Ideation-Chinese Version (BSI-CV) Score | baseline, immediately post-treatment and 2-week, 4-week and 8-week post-treatment
  BSI-CV is a self-reported questionnaire with 19 items. Each item is rated on a 3 point scale from 0 to 2. Scores range from 0 to 48. Total score Scores of 0 - 16 indicate low risk for suicide and scores of 16 or greater indicate higher risk for suicide.
Change in the Hamilton Anxiety Scale (HAMA) Score | baseline, immediately post-treatment and 2-week, 4-week and 8-week post-treatment
  HAMD total score comprises a sum of the 14 individual item scores. Each item is rated on a 5 point scale from 0 to 4. The Total Score can range from 0 to 56, and higher scores indicate a greater degree of anxiety.
Change From Baseline Functional Connectivity to Immediately Post-treatment | baseline、immediately post treatment and 4-week post-treatment
  The change in resting state fMRI functional connectivity of the pgACC to the default mode network and within the default mode network will be assessed.

OTHER OUTCOMES:
Change in a Neuropsychological Test Battery from Baseline to immediately post-treatment | Pre-treatment to immediately post-treatment
  The Perceived Deficits Questionnaire - Depression (PDQ-D) is a brief patient-rated scale to assess subjective cognitive dysfunction in people with depression. The PDQ-D is a 20-item questionnaire and the total score ranger from 0 to 80, and higher scores indicate a greater degree of cognitive impairment. THINC-it® is a brief screening tool designed to measure cognition and determine whether cognitive functioning is impaired. Users can complete the cognitive screening in only 10-15 minutes. THINC-it® includes 4 objective cognitive tests (adapted from choice reaction time, 1-back working memory task, symbol digit coding, and Trails-B) and a subjective cognitive questionnaire (PDQ-5).

CONTACTS AND LOCATIONS:
Locations (1):
- XijingH, Xi'an, Shaan'xi, China

IPD SHARING:
Plan to Share IPD: No
After completion of the trial and publication of the relevant paper, the corresponding author can be contacted for individual participant data.

REFERENCES:
- [Derived] Zheng K, Chen L, Wang H; DIRECT consortium; Li B, Chen B. Beyond depression symptoms: the default mode network as a predictor of antidepressant response. Npj Ment Health Res. 2026 Jan 16;5(1):2. doi: 10.1038/s44184-025-00182-2. PMID 41545765
- [Derived] Liu N, Zhao N, Tang N, Cai M, Zhang Y, Lv R, Zhang Y, Han T, Meng Y, Zang Y, Wang H. Safety and efficacy of individual target transcranial magnetic stimulation to stimulate the most negative correlate of DLPFC-pgACC in the treatment of major depressive disorder: study protocol of a double-blind, randomised controlled trial. BMJ Open. 2024 Nov 7;14(11):e081520. doi: 10.1136/bmjopen-2023-081520. PMID 39515856